CLINICAL TRIAL: NCT01370707
Title: A Randomized, Double-blind, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of CJ-30001 and CJ-30002 in Patients With Type 2 Diabetes and Inadequate Glycemic Control ; Phase III Study
Brief Title: A Study to Evaluate the Efficacy and Safety of CJ-30001 and CJ-30002 in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_VCM_301
Record Dates: First submitted 2011-06-02; First posted 2011-06-10 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- CJ-30001/CJ-30002 (Experimental)
  Interventions: Drug: CJ-30001/CJ-30002

INTERVENTIONS:
Drug: Metformin — 1000~1500mg/day, 24weeks
  Arms: Metformin
Drug: CJ-30001/CJ-30002 — 0.6/1500mg~0.9/1500mg/day, 24weeks
  Arms: CJ-30001/CJ-30002

SUMMARY:
The aim of this study is to evaluate the efficacy and safety fo CJ-30001/CJ-30002.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 Diabetes Mellitus
* 20~69 years old
* BMI < 30kg/m2
* HbA1c between 7% and 11%
* receiving no oral antihyperglycemic agent for more than seven days for at least 8 weeks
* Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

* Subjects with Type 1 Diabetes Mellitus
* FPG > 270mg/dL
* Subjects having insulin treatment
* Subjects with acute or chornic metaboic acidosis
* Subjects with cardiovascular disease
* Subjects with chronic GI disease
* Subjects with a history of substance or alchol abuse within 1 year
* Subjects with a history of hypersensitivity to biguanide or a-GI
* Subjects with hypopituitarism or hypocorticalism
* Subjects with cancer
* Subjects who take corticosteriods or plan to take corticosteroid
* AST and ALT > 2.5 times the upper limit of normal
* Creatinine level > 1.5mg/dL in male and 1.4mg/dL in female
* SBP > 150mmHg or DBP > 90mmHg
* Subjects who work the night shift
* Female subjects who are pregnant, breastfeeding or not using medically acceptable birth control
* Subjects who have participated in other study within 3 months
* Subjects judged to be unsuitable for this trial by investigator

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at week 24 | Baseline, week 24

SECONDARY OUTCOMES:
Change from baseline in HbA1c, FPG, insulin and GLP-1 at week 4, 8, 12, 18, 24 | Baseline, week 4, 8, 12, 18, 24
Change from baseline in 2hr PPG and postprandial insulin at week 24 | Baseline, week 24
Change from baseline in FPG and HbA1c according to HbA1c at baseline(7~8%,8~9%, 9~10%, 10~11%) | Baseline, week 4, 8, 12, 18, 24
Percentage of patients achieving HbA1c <7% at week 24 | week 24
Percentage of patients achieving HbA1c <6.5% at week 24 | week 24
Percentage of patients reaching FPG <126mg/dL at week 24 | week 24
Percentage of patients reaching 2hr PPG <200mg/dL at week 24 | week 24
Percentage of patients adjusting to the high dose | week 24
Percentage of withdrawing patients due to uncontrolled glucose | week 24
Change from baseline in serum lipid(T. cholesterol, HDL, LDL, TG) at week 24 | week 24
Glycemic variability | Baseline, week 8, 18, 24
  Glycemic variability is measured by M-value. M-value = ∑{|10*log(blood glucose/100)|3}/n+{Max(blood glucose)-Min(blood glucose)}/20, M<19: good, 19≤M<32: fair, 32≤M: poor

CONTACTS AND LOCATIONS:
Locations (21):
- South Korea (21):
  - Bucheon St. Mary's Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Bundang
  - Kyungpook University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - National Health Insurance Coporation Ilsan Hospital, Ilsan
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Inje University Pusan Baik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Eulji Medical Center, Seoul
  - Hallym University Medical Center(Gangdong), Seoul
  - Hallym University Medical Center(Gangnam), Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si